CLINICAL TRIAL: NCT02130024
Title: Development of New Geographic Atrophy in Patients With Neovascular (Wet) Age-related Macular Degeneration: a Comparison of Ranibizumab and Aflibercept
Brief Title: A Comparison of Ranibizumab and Aflibercept for the Development of Geographic Atrophy in (Wet) AMD Patients
Acronym: RIVAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFB002AAU17
Record Dates: First submitted 2014-03-27; First posted 2014-05-02 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2018-10

CONDITIONS: Age-Related Macular Degeneration
Keywords: Age-related macular degeneration; AMD; wet AMD; ranibizumab; aflibercept; geographic atrophy; inject and extend
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy | interventions — Ranibizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant
Masking Description: Investigators were not masked. The patients, the BCVA assessors, and the Central Reading Center (who set the treatment intervals) were masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ranibizumab 0.5 mg (Experimental): 3 monthly loading doses (Baseline, Week 4, and Week 8), followed by an individualised treatment and evaluation regimen according to disease activity [treat and extend]
  Interventions: Drug: Ranibizumab 0.5 mg
- Aflibercept 2.0 mg (Active Comparator): 3 monthly loading doses (Baseline, Week 4, and Week 8), followed by an individualised treatment and evaluation regimen according to disease activity [treat and extend]
  Interventions: Drug: Aflibercept 2.0 mg

INTERVENTIONS:
Drug: Ranibizumab 0.5 mg — Administered as an intravitreal injection
  Other Names: Lucentis
  Arms: Ranibizumab 0.5 mg
Drug: Aflibercept 2.0 mg — Administered as an intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept 2.0 mg

SUMMARY:
The purpose of this study was to compare the development of new geographic atrophy in patients with wet Age-related Macular Degeneration (AMD) when treated with either ranibizumab or aflibercept over 24 months. Geographic atrophy is an advanced form of AMD that can result in the progressive and irreversible loss of visual function over time.

DETAILED DESCRIPTION:
In each arm, patients underwent three monthly loading doses (at Baseline, Week 4, and Week 8). From Week 8, after the patient had received their third injection of study treatment, the visit intervals were determined by the patient's disease activity. If any of the protocol-specified signs of disease activity were present in the study eye, the subsequent injection visit interval was kept at 4 weeks. If none of the signs were present, the subsequent injection interval was extended by 2-week increments up until a maximum of 12-weekly intervals was reached. If there were any signs of disease activity in the study eye, the treatment interval was reduced as specified in the protocol. The planned individual duration of study participation was 24 months.

ELIGIBILITY:
Inclusion criteria:

- Written informed consent.

Inclusion criteria specific to the study eye:

* Diagnosis of active subfoveal Choroidal Neovascularisation (CNV) secondary to wet Age-related Macular Degeneration (AMD);
* Best Corrected Visual Acuity (BCVA) score of 23 letters or more as measured by 3-metre Early Treatment Diabetic Retinopathy Study (ETDRS)-like charts.

Exclusion criteria:

* Pregnant, nursing, or at risk of becoming pregnant during the study;
* Inability to comply with the study or follow-up procedures;
* Recent (3 months) stroke or myocardial infarction; uncontrolled hypertension; hypersensitivity to the study treatments or to fluorescein;
* In either eye: active periocular or ocular infection or inflammation; iris neovascularisation; uncontrolled or neovascular glaucoma; or one or more patch of geographic atrophy (GA) as specified in the protocol.

Exclusion criteria specific to the study eye:

* Prior or current treatment with anti-angiogenic drugs or corticosteroids;
* Other eye conditions as specified in the protocol;
* Any intraocular procedure carried out within 2 months before baseline or anticipated within 6 months following baseline.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (21):
- Australia (21):
  - Novartis Investigative Site, Albury, New South Wales
  - Novartis Investigative Site, Brookvale, New South Wales
  - Novartis Investigative Site, Chatswood, New South Wales
  - Novartis Investigative Site, Hurtsville, New South Wales
  - Novartis Investigative Site, Mona Vale, New South Wales
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Strathfield, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Sydney, NSW 2000
  - Novartis Investigative Site, Caboolture, Queensland
  - Novartis Investigative Site, Redcliffe, Queensland
  - Novartis Investigative Site, South Brisbane, Queensland
  - Novartis Investigative Site, Southport, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, South Launceston, Tasmania
  - Novartis Investigative Site, Clayton, Victoria
  - Novartis Investigative Site, Malvern, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Subiaco, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li E, Donati S, Lindsley KB, Krzystolik MG, Virgili G. Treatment regimens for administration of anti-vascular endothelial growth factor agents for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 May 5;5(5):CD012208. doi: 10.1002/14651858.CD012208.pub2. PMID 32374423
- [Derived] Gillies MC, Hunyor AP, Arnold JJ, Guymer RH, Wolf S, Ng P, Pecheur FL, McAllister IL. Effect of Ranibizumab and Aflibercept on Best-Corrected Visual Acuity in Treat-and-Extend for Neovascular Age-Related Macular Degeneration: A Randomized Clinical Trial. JAMA Ophthalmol. 2019 Apr 1;137(4):372-379. doi: 10.1001/jamaophthalmol.2018.6776. PMID 30676617

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited and enrolled from 24 sites located in Australia.
Pre-assignment Details: This reporting group includes all patients randomized to treatment.
Period: Overall Study
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Started | 142 | 139
Safety Set | 141 (One randomized patient did not receive treatment) | 139
Full Analysis Set (FAS) | 141 | 137 (2 patients had no post Baseline geographic atrophy (GA) data)
Completed | 117 | 108
Not Completed | 25 | 31
Not completed — Adverse Event | 10 | 11
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Deviation | 4 | 0
Not completed — Site Administration Problems | 1 | 0
Not completed — Subject Withdrew Consent | 6 | 14

BASELINE CHARACTERISTICS:
Population: All patients randomized to treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg | Total
Number analyzed (Participants) | 142 | 139 | 281
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.6 (8.5) | 78.7 (7.45) | 77.7 (8.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 76 | 148
  Male | 70 | 63 | 133
Race/Ethnicity, Customized [Number; unit: participants] — Predominant race
  participants
    Caucasian | 132 | 130 | 262
    Black African | 0 | 1 | 1
    Asian | 8 | 7 | 15
    Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Square-root Area of Geographic Atrophy (GA) From Baseline to Month 24
Description: Multimodal images of the eye were obtained by trained study site personnel and forwarded to an independent Central Reading Center, where the area of GA was measured. Area was treated as zero if GA was reported as absent (Overall determination of GA presence). Mean change from baseline in GA area was reported in square root-transformed data (mm). One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Month 24
Population: All randomized patients with at least one post-baseline efficacy value for the primary endpoint (FAS). Following the intent-to-treat principle, patients were analyzed according to the treatment regimen they were assigned to at randomization, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
mm
  Baseline: number analyzed (Participants) | 140 | 137
  Baseline | 0.024 (0.0988) | 0.050 (0.2345)
  Change from Baseline at Month 24: number analyzed (Participants) | 113 | 106
  Change from Baseline at Month 24 | 0.363 (0.7105) | 0.285 (0.5392)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Test type: Other; p = 0.236, Mixed Models Analysis; Fixed effects: Baseline GA area, treatment, visit, treatment by visit. Random effect: Subject; Treatment Effect = 0.08, 95% CI 2-sided [-0.05 to 0.21]

2. Secondary Outcome: Mean Change in Square-root Area of Geographic Atrophy From Baseline to Month 12
Description: as for outcome 1
Time Frame: Baseline, Month 12
Population: FAS. Following the intent-to-treat principle, patients were analyzed according to the treatment regimen they were assigned to at randomization, with no imputation for missing data.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
mm
  Baseline: number analyzed (Participants) | 140 | 137
  Baseline | 0.024 (0.0988) | 0.050 (0.2345)
  Change from Baseline at Month 12: number analyzed (Participants) | 125 | 120
  Change from Baseline at Month 12 | 0.155 (0.4272) | 0.145 (0.3179)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Test type: Other; p = 0.769, Mixed Models Analysis; Fixed effects: Baseline GA area, treatment, visit, treatment by visit. Random effect: Subject; Treatment Effect = 0.02, 95% CI 2-sided [-0.11 to 0.15]

3. Secondary Outcome: Percentage of Patients With Newly Developed Geographic Atrophy During the Overall 24 Months of the Study
Description: Multimodal images of the eye were obtained by trained study site personnel and forwarded to an independent Central Reading Center. A patient was considered to have developed new GA if they did not have any GA at the start of the study period and were subsequently diagnosed with GA during the study period (diagnosis of GA change from "No" to "Yes)." The analysis of new GA development was restricted to only those subjects without GA reported at baseline. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
percentage of patients
  Baseline to Month 12: number analyzed (Participants) | 125 | 118
  Baseline to Month 12 | 17.6 | 20.3
  Month 12 to Month 24: number analyzed (Participants) | 93 | 83
  Month 12 to Month 24 | 15.1 | 7.2
  Baseline to Month 24: number analyzed (Participants) | 125 | 118
  Baseline to Month 24 | 28.8 | 25.4
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 12 Analysis; Test type: Other; p = 0.586, Regression, Logistic; Includes treatment as factor. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 0.84, 95% CI 2-sided [0.44 to 1.59] — Odds ratio of 'Newly Developed GA (Yes)' at between the two treatment groups at study visit
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Month 12 to Month 24 Analysis; Test type: Other; p = 0.110, Regression, Logistic; Includes treatment as factor. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 2.27, 95% CI 2-sided [0.83 to 6.22] — Odds ratio of 'Newly Developed GA (Yes)' at between the two treatment groups at study visit
Statistical Analysis 3: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 24 Analysis; Test type: Other; p = 0.554, Regression, Logistic; Includes treatment as factor. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 1.19, 95% CI 2-sided [0.67 to 2.09]

4. Secondary Outcome: Mean Number of Intravitreal Injections From Baseline to Month 12 and to Month 24
Description: The number of intravitreal injections was calculated. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: injections
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
injections
  Baseline to Month 12 | 9.7 (2.78) | 9.7 (2.54)
  Month 12 to Month 24: number analyzed (Participants) | 127 | 121
  Month 12 to Month 24 | 8.9 (3.24) | 8.3 (3.56)
  Baseline to Month 24 | 17.7 (6.44) | 17.0 (6.3)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to <Month 12 Analysis; Test type: Other; p = 0.733, Negative Binomial Regression Model; Log (number of injections) = treatment + log (year of follow-up) (offset); Treatment Effect = 0.99, 95% CI 2-sided [0.95 to 1.04] — Treatment effect: Injection frequency (rate) ratio of Ranibizumab vs. Aflibercept
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 24 Analysis; Test type: Other; p = 0.745, Negative Binomial Regression Model; Log (number of injections) = treatment + log (year of follow-up) (offset); Treatment Effect = 1.01, 95% CI 2-sided [0.95 to 1.08] — Treatment effect: Injection frequency (rate) ratio of Ranibizumab vs. Aflibercept

5. Secondary Outcome: Mean Change in Best Corrected Visual Acuity (BCVA) From Baseline to Month 12 and to Month 24
Description: Visual acuity was assessed with spectacles or other visual corrective devices in place using logMAR charts and recorded in number of letters correctly identified. BCVA change was defined as a change in letters correctly identified from the baseline assessment. A positive change value indicates an improvement in visual acuity, while a negative change value indicates a worsening. One eye (study eye) contributed to the analysis
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
letters
  Baseline | 65.3 (15.10) | 65.1 (12.53)
  Change from Baseline at Month 12: number analyzed (Participants) | 127 | 121
  Change from Baseline at Month 12 | 6.9 (12.25) | 5.2 (12.83)
  Change from Baseline at Month 24: number analyzed (Participants) | 117 | 108
  Change from Baseline at Month 24 | 6.5 (14.38) | 5.3 (13.33)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 12 Analysis; Test type: Other; p = 0.079, Mixed Models Analysis; Fixed effects: Baseline BCVA, treatment, visit, and treatment by visit. Random effect: Subject. Response variable: Change from baseline in BCVA; Treatment Effect = 2.32, 95% CI 2-sided [-0.27 to 4.92] — Treatment Effect: Ranibizumab minus Aflibercept
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 24 Analysis; Test type: Other; p = 0.151, Mixed Models Analysis; [statistical method as in outcome 5, analysis 1]; Treatment Effect = 1.95, 95% CI 2-sided [-0.71 to 4.61] — Treatment Effect: Ranibizumab minus Aflibercept

6. Secondary Outcome: Mean Change in Central Subfield Foveal Thickness (CSFT) From Baseline to Month 12 and to Month 24
Description: CSFT (the average retinal thickness of the circular area within 1 millimeter diameter around the foveal center) was assessed using Optical Coherence Tomography (OCT) and measured in micrometers. A negative change value indicates an improvement, while a positive change value indicates a worsening. One eye (study eye) contributed to the analysis
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
micrometers
  Baseline | 468.2 (150.82) | 483.5 (168.05)
  Change from Baseline at Month 12: number analyzed (Participants) | 127 | 120
  Change from Baseline at Month 12 | -147.2 (128.38) | -171.6 (150.12)
  Change from Baseline at Month 24: number analyzed (Participants) | 117 | 108
  Change from Baseline at Month 24 | -151.3 (133.37) | -181.7 (155.48)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 12 Analysis; Test type: Other; p = 0.294, Mixed Models Analysis; Fixed effects: Baseline CSFT, treatment, visit, and treatment by visit. Random effect: Subject. Response variable: Change from baseline in CSFT; Treatment Effect = 10.12, 95% CI 2-sided [-8.82 to 29.06] — Treatment Effect: Ranibizumab minus Aflibercept
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 24 Analysis; Test type: Other; p = 0.225, Mixed Models Analysis; [statistical method as in outcome 6, analysis 1]; Treatment Effect = 11.86, 95% CI 2-sided [-7.35 to 31.07] — Treatment Effect: Ranibizumab minus Aflibercept

7. Secondary Outcome: Percentage of Patients Showing no Intraretinal Fluid (IRF)/Subretinal Fluid (SRF)
Description: Intraretinal fluid and subretinal fluid was assessed using Optical Coherence Tomography (OCT) and recorded as Present/Absent. One eye (study eye) contributed to the analysis.
Time Frame: Month 2, Month 12, Month 24
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
percentage of patients
  Month 2: number analyzed (Participants) | 137 | 137
  Month 2 | 56.9 | 61.3
  Month 12: number analyzed (Participants) | 127 | 121
  Month 12 | 55.9 | 63.6
  Month 24: number analyzed (Participants) | 117 | 109
  Month 24 | 57.3 | 60.6
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Month 2 Analysis; Test type: Other; p = 0.461, Regression, Logistic; Includes treatment as factor. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 0.83, 95% CI 2-sided [0.51 to 1.35] — Odds ratio of no IRF/SRF present between the two treatment groups at study visit
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Month 12 Analysis; Test type: Other; p = 0.215, Regression, Logistic; Includes treatment as factor. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.44 to 1.21] — Odds ratio of no IRF/SRF present between the two treatment groups at study visit
Statistical Analysis 3: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Month 24 Analysis; Test type: Other; p = 0.616, Regression, Logistic; Includes treatment as factor. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.51 to 1.48] — Odds ratio of no IRF/SRF present between the two treatment groups at study visit

8. Secondary Outcome: Percentage of Patients Showing Greater Than and Equal to 15 Letters Gain for BCVA From Baseline to Month 12 and to Month 24
Description: Visual acuity was assessed with spectacles or other visual corrective devices in place using logMAR charts and recorded in number of letters correctly identified. A gain in letters correctly identified indicates an improvement in visual acuity, while a loss indicates a worsening. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
percentage of patients
  Change from Baseline at Month 12: number analyzed (Participants) | 127 | 121
  Change from Baseline at Month 12 | 22.0 | 20.7
  Change from Baseline at Month 24: number analyzed (Participants) | 117 | 108
  Change from Baseline at Month 24 | 24.8 | 18.5
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 12 Analysis; Test type: Other; p = 0.891, Regression, Logistic; Includes treatment as factor and baseline BCVA as covariate. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.53 to 2.08] — Odds ratio of BCVA change from baseline ≥15 letters between the two treatment groups at study visit
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 24 Analysis; Test type: Other; p = 0.206, Regression, Logistic; Includes treatment as factor and baseline BCVA as covariate. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.77 to 3.35] — Odds ratio of BCVA change from baseline ≥15 letters between the two treatment groups at study visit

9. Secondary Outcome: Percentage of Patients Showing Less Than and Equal to 15 Letters Loss for BCVA From Baseline to Month 12 and to Month 24
Description: as for outcome 8
Time Frame: Baseline, Month 12, Month 24
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
percentage of patients
  Change from Baseline at Month 12: number analyzed (Participants) | 127 | 121
  Change from Baseline at Month 12 | 96.9 | 95.0
  Change from Baseline at Month 24: number analyzed (Participants) | 117 | 108
  Change from Baseline at Month 24 | 94.0 | 94.4
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 12 Analysis; Test type: Other; p = 0.460, Regression, Logistic; Includes treatment as factor and baseline BCVA as covariate. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 1.63, 95% CI 2-sided [0.45 to 5.93] — Odds ratio of BCVA change from baseline ≥ -15 letters between the two treatment groups at study visit
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Month 24 Analysis; Test type: Other; p = 0.913, Regression, Logistic; Includes treatment as factor and baseline BCVA as covariate. Model: log(p/1-p) =Treatment; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.30 to 2.90] — Odds ratio of BCVA change from baseline ≥ -15 letters between the two treatment groups at study visit

10. Secondary Outcome: Mean Number of Times a Patient Needed to Return to Monthly Intravitreal Injections Over 24 Months
Description: The number of times the patient returned to a monthly injection interval (from an extended interval) at least once during the 24-month study was calculated. One eye (study eye) contributed to the analysis.
Time Frame: Month 24
Population: FAS. Following the intent-to-treat principle, patients were analyzed according to the treatment regimen they were assigned to at randomization, with no imputation for missing data. Descriptive statistics only.
Measure: Mean (Standard Deviation); unit: occurrences
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 134 | 134
occurrences | 2.3 (1.28) | 2.3 (1.15)

11. Secondary Outcome: Mean Change in Vascular Endothelial Growth Factor (VEGF) Plasma Concentration From Baseline to 7 Days After the Second and 7 Days After the Third Mandated Intravitreal Injection of Treatment
Description: Blood for VEGF plasma concentration analysis was collected at Baseline and again at 7 days after the injection at Week 4 and 7 days after the injection at Week 8.
Time Frame: Baseline, Week 5, Week 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: picogram/milliliter (pg/mL)
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 137
picogram/milliliter (pg/mL)
  Baseline: number analyzed (Participants) | 139 | 137
  Baseline | 44.29 (43.369) | 41.88 (35.236)
  Change from Baseline at Week 5: number analyzed (Participants) | 130 | 135
  Change from Baseline at Week 5 | -0.48 (30.299) | -26.37 (36.220)
  Change from Baseline at Week 9: number analyzed (Participants) | 129 | 131
  Change from Baseline at Week 9 | 0.48 (35.125) | -25.14 (32.525)
Statistical Analysis 1: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Week 5 Analysis; Test type: Other; p < 0.001, Mixed Models Analysis; Fixed: BL Plasma VEGF, treatment, visit, and treatment by visit. Random effect: Subject. Response variable: Change from BL in Plasma VEGF; Treatment Effect = 27.20, 95% CI 2-sided [21.44 to 32.95] — Treatment Effect: Ranibizumab minus Aflibercept
Statistical Analysis 2: Comparison: Ranibizumab 0.5 mg vs Aflibercept 2.0 mg; Baseline to Week 9 Analysis; Test type: Other; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 11, analysis 1]; Treatment Effect = 28.88, 95% CI 2-sided [23.08 to 34.68] — Treatment Effect: Ranibizumab minus Aflibercept

12. Secondary Outcome: Percentage of Patients With Change in Retinal Nerve Fibre Thickness From Baseline to Month 12 and Month 24
Description: Retinal nerve fibre thickness was assessed using Optical Coherence Tomography (OCT) and measured in micrometers. A negative change in value (i.e. thinner nerve fibre) indicates nerve damage. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Month 12, Month 24
Population: Safety Set. All patients who received at least one application of study treatment and had at least one post-baseline safety assessment, as treated. Descriptive statistics only.
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 139
percentage of patients
  Month 12: Decrease from Baseline: number analyzed (Participants) | 122 | 111
  Month 12: Decrease from Baseline | 2.5 | 2.7
  Month 12: No Change from Baseline: number analyzed (Participants) | 122 | 111
  Month 12: No Change from Baseline | 96.7 | 97.3
  Month 12: Increase from Baseline: number analyzed (Participants) | 122 | 111
  Month 12: Increase from Baseline | 0.8 | 0
  Month 24: Decrease from Baseline: number analyzed (Participants) | 110 | 97
  Month 24: Decrease from Baseline | 3.6 | 1.0
  Month 24: No Change from Baseline: number analyzed (Participants) | 110 | 97
  Month 24: No Change from Baseline | 96.4 | 97.9
  Month 24: Increase from Baseline: number analyzed (Participants) | 110 | 97
  Month 24: Increase from Baseline | 0 | 1.0

13. Secondary Outcome: Percentage of Patients With Ocular Inflammation at Baseline and 7 Days Post-injection Following 3rd Mandated Intravitreal Injection - Anterior Chamber Cells
Description: Anterior cell grade was assessed by the Investigator during slit lamp examination and graded on a 5-point scale: Grade 0=0 cells; Grade 1=1 to 10 cells; Grade 2=11 to 20 cells; Grade 3=21 to 50 cells; Grade 4=>50 cells. The presence of blood cells (red and white) in the anterior chamber of the eye (the fluid-filled space inside the eye between the iris and the cornea's innermost surface) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 9
Population: as for outcome 12
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 138
percentage of patients
  Baseline: Grade 0: number analyzed (Participants) | 136 | 135
  Baseline: Grade 0 | 99.3 | 98.5
  Baseline: Grade 1+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 1+ | 0.7 | 1.5
  Baseline: Grade 2+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 2+ | 0 | 0
  Baseline: Grade 3+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 3+ | 0 | 0
  Baseline: Grade 4+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 4+ | 0 | 0
  Week 9: Grade 0: number analyzed (Participants) | 123 | 123
  Week 9: Grade 0 | 95.1 | 92.7
  Week 9: Grade 1+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 1+ | 4.9 | 7.3
  Week 9: Grade 2+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 2+ | 0 | 0
  Week 9: Grade 3+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 3+ | 0 | 0
  Week 9: Grade 4+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 4+ | 0 | 0

14. Secondary Outcome: Percentage of Patients With Ocular Inflammation at Baseline and 7 Days Post-injection Following 3rd Mandated Intravitreal Injection - Anterior Chamber Flare
Description: Anterior chamber flare was assessed by the investigator during slit lamp examination and graded on a 5-point scale, with 0 = none; 1 = mild (trace to clearly noticeable, visible); 2 = moderate; 3 = marked; and 4 = severe. The presence of flare (increased protein levels) in the anterior chamber of the eye (the fluid-filled space inside the eye between the iris and the cornea's innermost surface) is a sign of intraocular inflammation. A score of 0 indicates an absence of inflammation. Proportion of patients is reported as a percentage. One eye (study eye) contributed to the analysis.
Time Frame: Baseline, Week 9
Population: as for outcome 12
Measure: Number; unit: percentage of patients
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
Number analyzed (Participants) | 141 | 138
percentage of patients
  Baseline: Grade 0: number analyzed (Participants) | 136 | 135
  Baseline: Grade 0 | 97.8 | 99.3
  Baseline: Grade 1+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 1+ | 2.2 | 0.7
  Baseline: Grade 2+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 2+ | 0 | 0
  Baseline: Grade 3+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 3+ | 0 | 0
  Baseline: Grade 4+: number analyzed (Participants) | 136 | 135
  Baseline: Grade 4+ | 0 | 0
  Week 9: Grade 0: number analyzed (Participants) | 123 | 123
  Week 9: Grade 0 | 94.3 | 92.7
  Week 9: Grade 1+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 1+ | 5.7 | 7.3
  Week 9: Grade 2+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 2+ | 0 | 0
  Week 9: Grade 3+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 3+ | 0 | 0
  Week 9: Grade 4+: number analyzed (Participants) | 123 | 123
  Week 9: Grade 4+ | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the individual's participation in the study (approximately 24 months).
Description: This analysis population includes all patients who received at least one application of study treatment and had at least one post-baseline safety assessment (Safety Analysis Set).
Arm/Group | Ranibizumab 0.5 mg | Aflibercept 2.0 mg
All-Cause Mortality (participants affected / at risk) | 3/141 | 6/139
Serious Adverse Events (participants affected / at risk) | 50/141 | 58/139
Other Adverse Events (participants affected / at risk) | 122/141 | 123/139
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=141) | Aflibercept 2.0 mg (N=139)
Anaemia (Non-ocular) (Blood and lymphatic system disorders) | 0 | 1
Iron deficiency anaemia (Non-ocular) (Blood and lymphatic system disorders) | 1 | 1
Platelet dysfunction (Non-ocular) (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Non-ocular) (Cardiac disorders) | 1 | 1
Aortic valve incompetence (Non-ocular) (Cardiac disorders) | 1 | 0
Atrial fibrillation (Non-ocular) (Cardiac disorders) | 7 | 0
Atrioventricular block complete (Non-ocular) (Cardiac disorders) | 0 | 1
Cardiac arrest (Non-ocular) (Cardiac disorders) | 0 | 1
Cardiac failure (Non-ocular) (Cardiac disorders) | 1 | 1
Cardiac failure chronic (Non-ocular) (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Non-ocular) (Cardiac disorders) | 1 | 0
Coronary artery disease (Non-ocular) (Cardiac disorders) | 0 | 1
Left ventricular failure (Non-ocular) (Cardiac disorders) | 0 | 2
Myocardial infarction (Non-ocular) (Cardiac disorders) | 1 | 0
Palpitations (Non-ocular) (Cardiac disorders) | 1 | 1
Tachycardia (Non-ocular) (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Non-ocular) (Cardiac disorders) | 0 | 1
Meniere's disease (Non-ocular) (Ear and labyrinth disorders) | 1 | 0
Retinal artery embolism (Right eye) (Eye disorders) | 1 | 0
Retinal artery occlusion (Right eye) (Eye disorders) | 1 | 0
Retinal detachment (Left eye) (Eye disorders) | 0 | 2
Constipation (Non-ocular) (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Non-ocular) (Gastrointestinal disorders) | 0 | 1
Diverticulum (Non-ocular) (Gastrointestinal disorders) | 0 | 1
Gastritis (Non-ocular) (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Non-ocular) (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Non-ocular) (Gastrointestinal disorders) | 0 | 1
Localised intraabdominal fluid collection (Non-ocular) (Gastrointestinal disorders) | 0 | 1
Nausea (Non-ocular) (Gastrointestinal disorders) | 1 | 1
Oesophageal food impaction (Non-ocular) (Gastrointestinal disorders) | 1 | 1
Peritoneal adhesions (Non-ocular) (Gastrointestinal disorders) | 1 | 0
Pharyngo-oesophageal diverticulum (Non-ocular) (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Non-ocular) (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Non-ocular) (Gastrointestinal disorders) | 1 | 0
Volvulus (Non-ocular) (Gastrointestinal disorders) | 1 | 0
Vomiting (Non-ocular) (Gastrointestinal disorders) | 1 | 0
Chest pain (Non-ocular) (General disorders) | 3 | 2
Condition aggravated (Non-ocular) (General disorders) | 0 | 2
Death (Non-ocular) (General disorders) | 1 | 1
Disease progression (Non-ocular) (General disorders) | 0 | 1
General physical health deterioration (Non-ocular) (General disorders) | 0 | 1
Hernia (Non-ocular) (General disorders) | 0 | 1
Pyrexia (Non-ocular) (General disorders) | 0 | 1
Bile duct stone (Non-ocular) (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Non-ocular) (Hepatobiliary disorders) | 1 | 0
Blastocystis infection (Non-ocular) (Infections and infestations) | 0 | 1
Cellulitis (Non-ocular) (Infections and infestations) | 1 | 2
Clostridium difficile colitis (Non-ocular) (Infections and infestations) | 1 | 0
Cystitis (Non-ocular) (Infections and infestations) | 0 | 1
Endophthalmitis (Left eye) (Infections and infestations) | 0 | 1
Endophthalmitis (Right eye) (Infections and infestations) | 0 | 1
Escherichia infection (Non-ocular) (Infections and infestations) | 1 | 0
Gallbladder empyema (Non-ocular) (Infections and infestations) | 1 | 0
Gastroenteritis (Non-ocular) (Infections and infestations) | 1 | 1
Gastroenteritis viral (Non-ocular) (Infections and infestations) | 0 | 1
Herpes zoster (Non-ocular) (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Non-ocular) (Infections and infestations) | 2 | 0
Influenza (Non-ocular) (Infections and infestations) | 1 | 0
Localised infection (Non-ocular) (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Non-ocular) (Infections and infestations) | 2 | 0
Onychomycosis (Non-ocular) (Infections and infestations) | 1 | 0
Pneumonia (Non-ocular) (Infections and infestations) | 4 | 4
Pneumonia bacterial (Non-ocular) (Infections and infestations) | 1 | 0
Rhinovirus infection (Non-ocular) (Infections and infestations) | 0 | 1
Sepsis (Non-ocular) (Infections and infestations) | 1 | 1
Septic shock (Non-ocular) (Infections and infestations) | 1 | 0
Subcutaneous abscess (Non-ocular) (Infections and infestations) | 0 | 1
Urinary tract infection (Non-ocular) (Infections and infestations) | 2 | 4
Urinary tract infection bacterial (Non-ocular) (Infections and infestations) | 0 | 1
Ankle fracture (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Back injury (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Cataract traumatic (Right eye) (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Fall (Non-ocular) (Injury, poisoning and procedural complications) | 3 | 1
Femoral neck fracture (Non-ocular) (Injury, poisoning and procedural complications) | 3 | 2
Femur fracture (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 2
Fibula fracture (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Forearm fracture (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 1
Spinal column injury (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Non-ocular) (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Non-ocular) (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Non-ocular) (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Non-ocular) (Metabolism and nutrition disorders) | 0 | 2
Malnutrition (Non-ocular) (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Non-ocular) (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Non-ocular) (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc space narrowing (Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Non-ocular) (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Non-ocular) (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Non-ocular) (Musculoskeletal and connective tissue disorders) | 2 | 1
Spinal column stenosis (Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 0
Adrenal gland cancer (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angioimmunoblastic T-cell lymphoma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 2
Benign ovarian tumour (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign uterine neoplasm (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer recurrent (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder neoplasm (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal carcinoma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant melanoma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant neoplasm progression (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mesothelioma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloproliferative disorder (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal cancer metastatic (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Sinonasal papilloma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Tonsil cancer (Non-ocular) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Non-ocular) (Nervous system disorders) | 1 | 0
Aphasia (Non-ocular) (Nervous system disorders) | 3 | 0
Basal ganglia haemorrhage (Non-ocular) (Nervous system disorders) | 1 | 0
Cerebral artery thrombosis (Non-ocular) (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Non-ocular) (Nervous system disorders) | 1 | 3
Dementia (Non-ocular) (Nervous system disorders) | 1 | 0
Dizziness (Non-ocular) (Nervous system disorders) | 1 | 0
Dysarthria (Non-ocular) (Nervous system disorders) | 0 | 1
Ischaemic stroke (Non-ocular) (Nervous system disorders) | 1 | 0
Lacunar infarction (Non-ocular) (Nervous system disorders) | 1 | 0
Neuralgia (Non-ocular) (Nervous system disorders) | 0 | 1
Presyncope (Non-ocular) (Nervous system disorders) | 1 | 0
Subarachnoid haemorrhage (Non-ocular) (Nervous system disorders) | 1 | 0
Syncope (Non-ocular) (Nervous system disorders) | 3 | 2
Transient ischaemic attack (Non-ocular) (Nervous system disorders) | 2 | 1
Delirium (Non-ocular) (Psychiatric disorders) | 1 | 1
Depression (Non-ocular) (Psychiatric disorders) | 0 | 1
Haematuria (Non-ocular) (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Non-ocular) (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Non-ocular) (Renal and urinary disorders) | 0 | 1
Renal failure acute (Non-ocular) (Renal and urinary disorders) | 3 | 2
Urethral haemorrhage (Non-ocular) (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Non-ocular) (Renal and urinary disorders) | 0 | 1
Urinary retention (Non-ocular) (Renal and urinary disorders) | 0 | 2
Ovarian cyst (Non-ocular) (Reproductive system and breast disorders) | 1 | 0
Prostatomegaly (Non-ocular) (Reproductive system and breast disorders) | 0 | 1
Uterovaginal prolapse (Non-ocular) (Reproductive system and breast disorders) | 0 | 1
Vaginal ulceration (Non-ocular) (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Open reduction of fracture (Non-ocular) (Surgical and medical procedures) | 1 | 0
Aortic dilatation (Non-ocular) (Vascular disorders) | 1 | 0
Aortic embolus (Non-ocular) (Vascular disorders) | 1 | 0
Aortic stenosis (Non-ocular) (Vascular disorders) | 1 | 0
Hypertension (Non-ocular) (Vascular disorders) | 1 | 0
Hypotension (Non-ocular) (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5 mg (N=141) | Aflibercept 2.0 mg (N=139)
Anaemia (Non-ocular) (Blood and lymphatic system disorders) | 4 | 4
Angina pectoris (Non-ocular) (Cardiac disorders) | 1 | 3
Atrial fibrillation (Non-ocular) (Cardiac disorders) | 3 | 4
Bundle branch block left (Non-ocular) (Cardiac disorders) | 0 | 3
Tachycardia (Non-ocular) (Cardiac disorders) | 2 | 3
Vertigo (Non-ocular) (Ear and labyrinth disorders) | 0 | 5
Age-related macular degeneration (Left eye) (Eye disorders) | 6 | 8
Age-related macular degeneration (Right eye) (Eye disorders) | 10 | 14
Blepharitis (Both eyes) (Eye disorders) | 3 | 2
Cataract (Both eyes) (Eye disorders) | 1 | 3
Cataract (Left eye) (Eye disorders) | 3 | 14
Cataract (Right eye) (Eye disorders) | 6 | 8
Chalazion (Left eye) (Eye disorders) | 2 | 4
Chalazion (Right eye) (Eye disorders) | 1 | 3
Choroidal neovascularisation (Left eye) (Eye disorders) | 2 | 3
Choroidal neovascularisation (Right eye) (Eye disorders) | 6 | 5
Conjunctival haemorrhage (Left eye) (Eye disorders) | 6 | 3
Dry eye (Both eyes) (Eye disorders) | 13 | 9
Dry eye (Left eye) (Eye disorders) | 1 | 3
Eye discharge (Both eyes) (Eye disorders) | 0 | 3
Eye discharge (Left eye) (Eye disorders) | 3 | 0
Eye discharge (Right eye) (Eye disorders) | 2 | 3
Eye irritation (Both eyes) (Eye disorders) | 2 | 3
Eye irritation (Left eye) (Eye disorders) | 5 | 3
Eye irritation (Right eye) (Eye disorders) | 2 | 4
Eye pain (Both eyes) (Eye disorders) | 6 | 0
Eye pain (Left eye) (Eye disorders) | 10 | 15
Eye pain (Right eye) (Eye disorders) | 14 | 13
Eye pruritus (Both eyes) (Eye disorders) | 1 | 4
Lacrimation increased (Both eyes) (Eye disorders) | 4 | 5
Lacrimation increased (Left eye) (Eye disorders) | 5 | 3
Lacrimation increased (Right eye) (Eye disorders) | 3 | 3
Macular degeneration (Right eye) (Eye disorders) | 3 | 3
Metamorphopsia (Left eye) (Eye disorders) | 1 | 3
Metamorphopsia (Right eye) (Eye disorders) | 0 | 3
Ocular hyperaemia (Left eye) (Eye disorders) | 3 | 7
Ocular hyperaemia (Right eye) (Eye disorders) | 4 | 4
Posterior capsule opacification (Right eye) (Eye disorders) | 2 | 4
Retinal haemorrhage (Left eye) (Eye disorders) | 3 | 5
Retinal haemorrhage (Right eye) (Eye disorders) | 5 | 3
Retinal pigment epithelial tear (Left eye) (Eye disorders) | 5 | 3
Vision blurred (Both eyes) (Eye disorders) | 4 | 1
Vision blurred (Left eye) (Eye disorders) | 2 | 5
Vision blurred (Right eye) (Eye disorders) | 3 | 6
Visual acuity reduced (Right eye) (Eye disorders) | 6 | 2
Vitreous detachment (Both eyes) (Eye disorders) | 4 | 2
Vitreous detachment (Left eye) (Eye disorders) | 3 | 12
Vitreous detachment (Right eye) (Eye disorders) | 2 | 11
Vitreous floaters (Both eyes) (Eye disorders) | 4 | 2
Vitreous floaters (Left eye) (Eye disorders) | 7 | 7
Vitreous floaters (Right eye) (Eye disorders) | 7 | 9
Abdominal pain (Non-ocular) (Gastrointestinal disorders) | 0 | 5
Constipation (Non-ocular) (Gastrointestinal disorders) | 6 | 13
Diarrhoea (Non-ocular) (Gastrointestinal disorders) | 7 | 5
Gastrooesophageal reflux disease (Non-ocular) (Gastrointestinal disorders) | 3 | 10
Nausea (Non-ocular) (Gastrointestinal disorders) | 12 | 6
Vomiting (Non-ocular) (Gastrointestinal disorders) | 4 | 5
Asthenia (Non-ocular) (General disorders) | 3 | 0
Chest pain (Non-ocular) (General disorders) | 4 | 4
Influenza like illness (Non-ocular) (General disorders) | 8 | 3
Malaise (Non-ocular) (General disorders) | 1 | 4
Oedema peripheral (Non-ocular) (General disorders) | 2 | 3
Pain (Right eye) (General disorders) | 0 | 3
Pyrexia (Non-ocular) (General disorders) | 4 | 2
Drug hypersensitivity (Both eyes) (Immune system disorders) | 3 | 0
Drug hypersensitivity (Non-ocular) (Immune system disorders) | 4 | 3
Seasonal allergy (Non-ocular) (Immune system disorders) | 6 | 1
Bronchitis (Non-ocular) (Infections and infestations) | 4 | 1
Cellulitis (Non-ocular) (Infections and infestations) | 0 | 3
Diverticulitis (Non-ocular) (Infections and infestations) | 3 | 1
Gastroenteritis (Non-ocular) (Infections and infestations) | 2 | 3
Herpes zoster (Non-ocular) (Infections and infestations) | 4 | 4
Influenza (Non-ocular) (Infections and infestations) | 11 | 6
Lower respiratory tract infection (Non-ocular) (Infections and infestations) | 11 | 6
Nasopharyngitis (Non-ocular) (Infections and infestations) | 15 | 8
Pneumonia (Non-ocular) (Infections and infestations) | 2 | 4
Sinusitis (Non-ocular) (Infections and infestations) | 1 | 3
Upper respiratory tract infection (Non-ocular) (Infections and infestations) | 8 | 11
Urinary tract infection (Non-ocular) (Infections and infestations) | 11 | 15
Contusion (Non-ocular) (Injury, poisoning and procedural complications) | 1 | 3
Corneal abrasion (Right eye) (Injury, poisoning and procedural complications) | 4 | 2
Fall (Non-ocular) (Injury, poisoning and procedural complications) | 11 | 15
Head injury (Non-ocular) (Injury, poisoning and procedural complications) | 0 | 3
Abdominal X-ray (Non-ocular) (Investigations) | 1 | 4
Angiogram (Non-ocular) (Investigations) | 4 | 3
Arteriogram coronary (Non-ocular) (Investigations) | 3 | 4
Biopsy (Non-ocular) (Investigations) | 0 | 4
Blood alkaline phosphatase increased (Non-ocular) (Investigations) | 1 | 3
Blood chloride decreased (Non-ocular) (Investigations) | 3 | 3
Blood cholesterol increased (Non-ocular) (Investigations) | 3 | 0
Blood creatinine increased (Non-ocular) (Investigations) | 1 | 4
Blood sodium decreased (Non-ocular) (Investigations) | 3 | 2
Blood urea increased (Non-ocular) (Investigations) | 2 | 4
C-reactive protein increased (Non-ocular) (Investigations) | 3 | 6
Chest X-ray (Non-ocular) (Investigations) | 14 | 20
Colonoscopy (Non-ocular) (Investigations) | 6 | 6
Computerised tomogram (Non-ocular) (Investigations) | 6 | 18
Computerised tomogram abdomen (Non-ocular) (Investigations) | 3 | 2
Computerised tomogram head (Non-ocular) (Investigations) | 11 | 11
Cystoscopy (Non-ocular) (Investigations) | 2 | 3
Echocardiogram (Non-ocular) (Investigations) | 9 | 13
Electrocardiogram (Non-ocular) (Investigations) | 7 | 5
Electrocardiogram ambulatory (Non-ocular) (Investigations) | 0 | 3
Full blood count (Non-ocular) (Investigations) | 3 | 1
Gamma-glutamyltransferase increased (Non-ocular) (Investigations) | 0 | 4
Glomerular filtration rate decreased (Non-ocular) (Investigations) | 2 | 3
Haematocrit decreased (Non-ocular) (Investigations) | 0 | 4
Haemoglobin decreased (Non-ocular) (Investigations) | 2 | 4
International normalised ratio increased (Non-ocular) (Investigations) | 1 | 3
Intraocular pressure increased (Left eye) (Investigations) | 1 | 3
Lymphocyte count decreased (Non-ocular) (Investigations) | 2 | 4
Neutrophil count increased (Non-ocular) (Investigations) | 2 | 5
Nuclear magnetic resonance imaging (Non-ocular) (Investigations) | 2 | 4
Nuclear magnetic resonance imaging brain (Non-ocular) (Investigations) | 5 | 3
Red blood cell count decreased (Non-ocular) (Investigations) | 0 | 3
Ultrasound Doppler (Non-ocular) (Investigations) | 5 | 4
Ultrasound abdomen (Non-ocular) (Investigations) | 1 | 3
Ultrasound kidney (Non-ocular) (Investigations) | 2 | 3
Weight decreased (Non-ocular) (Investigations) | 0 | 3
White blood cell count increased (Non-ocular) (Investigations) | 2 | 5
X-ray (Non-ocular) (Investigations) | 5 | 1
X-ray limb (Non-ocular) (Investigations) | 3 | 1
X-ray of pelvis and hip (Non-ocular) (Investigations) | 2 | 5
Hypercholesterolaemia (Non-ocular) (Metabolism and nutrition disorders) | 5 | 1
Hypokalaemia (Non-ocular) (Metabolism and nutrition disorders) | 3 | 4
Vitamin D deficiency (Non-ocular) (Metabolism and nutrition disorders) | 1 | 3
Arthralgia (Non-ocular) (Musculoskeletal and connective tissue disorders) | 6 | 7
Arthritis (Non-ocular) (Musculoskeletal and connective tissue disorders) | 4 | 2
Back pain (Non-ocular) (Musculoskeletal and connective tissue disorders) | 9 | 8
Muscular weakness (Non-ocular) (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Non-ocular) (Musculoskeletal and connective tissue disorders) | 5 | 1
Osteoarthritis (Non-ocular) (Musculoskeletal and connective tissue disorders) | 4 | 2
Osteoporosis (Non-ocular) (Musculoskeletal and connective tissue disorders) | 1 | 4
Pain in extremity (Non-ocular) (Musculoskeletal and connective tissue disorders) | 3 | 2
Dizziness (Non-ocular) (Nervous system disorders) | 5 | 7
Headache (Non-ocular) (Nervous system disorders) | 6 | 12
Lethargy (Non-ocular) (Nervous system disorders) | 3 | 3
Migraine (Non-ocular) (Nervous system disorders) | 3 | 0
Neuralgia (Non-ocular) (Nervous system disorders) | 3 | 1
Sciatica (Non-ocular) (Nervous system disorders) | 3 | 2
Anxiety (Non-ocular) (Psychiatric disorders) | 0 | 4
Delirium (Non-ocular) (Psychiatric disorders) | 3 | 2
Insomnia (Non-ocular) (Psychiatric disorders) | 1 | 7
Haematuria (Non-ocular) (Renal and urinary disorders) | 2 | 6
Renal cyst (Non-ocular) (Renal and urinary disorders) | 2 | 3
Renal impairment (Non-ocular) (Renal and urinary disorders) | 1 | 3
Urinary incontinence (Non-ocular) (Renal and urinary disorders) | 3 | 2
Asthma (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Dyspnoea (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Oropharyngeal pain (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Productive cough (Non-ocular) (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Rash (Non-ocular) (Skin and subcutaneous tissue disorders) | 4 | 6
Skin lesion (Non-ocular) (Skin and subcutaneous tissue disorders) | 3 | 0
Cancer surgery (Non-ocular) (Surgical and medical procedures) | 6 | 5
Cardiac pacemaker insertion (Non-ocular) (Surgical and medical procedures) | 1 | 3
Cataract operation (Left eye) (Surgical and medical procedures) | 4 | 11
Cataract operation (Right eye) (Surgical and medical procedures) | 10 | 7
Hip arthroplasty (Non-ocular) (Surgical and medical procedures) | 5 | 6
Inguinal hernia repair (Non-ocular) (Surgical and medical procedures) | 0 | 3
Intraocular lens implant (Right eye) (Surgical and medical procedures) | 2 | 4
Radiotherapy (Non-ocular) (Surgical and medical procedures) | 3 | 2
Skin neoplasm excision (Non-ocular) (Surgical and medical procedures) | 9 | 6
Transfusion (Non-ocular) (Surgical and medical procedures) | 3 | 0
Hypertension (Non-ocular) (Vascular disorders) | 8 | 12
Hypotension (Non-ocular) (Vascular disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2015-01-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT02130024/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/24/NCT02130024/SAP_001.pdf